CLINICAL TRIAL: NCT02182518
Title: Double-blind, Randomized, Parallel Trial to Evaluate the Clinical Efficacy and Safety of Epinastine 10 mg + Pseudoephedrine 120 mg SR, Twice a Day, Versus Epinastine 10 mg Alone, Twice a Day, in the Treatment of Outpatients With Perennial Allergic Rhinitis
Brief Title: Epinastine + Pseudoephedrine SR (Slow Release) Versus Epinastine Alone in Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 262.254
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — epinastine; Pseudoephedrine

ARMS (2):
- Epinastine + Pseudoephedrine (Experimental)
  Interventions: Drug: Epinastine; Drug: Pseudoephedrine; Drug: Placebo
- Epinastine (Experimental)
  Interventions: Drug: Epinastine; Drug: Placebo

INTERVENTIONS:
Drug: Epinastine
Drug: Pseudoephedrine
  Arms: Epinastine + Pseudoephedrine
Drug: Placebo — Placebo during run-in period

SUMMARY:
The aim of this trial is to evaluate the clinical efficacy and safety of Epinastine 10 mg + Pseudoephedrine 120 mg slow release (SR) administered twice a day, compared to Epinastine 10 mg alone administered twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients
* Over 12 years old
* Patients who have granted their written informed consent, personally or by a legal representative, to be part of the study and in accomplishment of the model of informed consent approved by the Ethic Committee of the institution
* Patients with an established diagnosis of allergic perennial rhinitis under the clinical criteria (allergic to one or more allergens)
* Patients with moderate or complete nasal blockage characterizes by ≥50 mm in the VAS for this parameter during visits 1 and 2
* Patients with positive (≥3 mm compared to the negative control) skin test ("Prick Test") to one or more of the following allergens:

  * Dermatophagoides pteronyssinus
  * Dermatophagoides farinae
  * Blomia tropicalis
  * Alternaria alternata
  * Cladosporium herbarum
  * Aspergillus fumigatus
  * Penicillium notatum
  * cat's fur
  * dog's fur

Exclusion Criteria:

* Pregnant or breast feeding women, or women without contraceptive method who:

  * are not in the postmenopausal period and/or
  * have not been submitted to bilateral tubal ligation or hysterectomy and/or
  * are not under one of the following contraceptive control:

    * oral contraceptive
    * IUD (intrauterine device)
    * diaphragm
* Patients unable to understand, accept or follow the protocol instructions
* History of serious adverse events with antihistamines
* Patients under treatment with calcium antagonists or other antihypertensive drugs
* Patients under treatment with digitalis
* Patients under treatment with MAO (monoamine oxidase) inhibitors
* Patients under treatment with sympathicomimetics
* Patients that have received any of the following drugs during the periods specified below, before visit 1:

  * Inhaled/Topics

    * short acting β2 agonists (12 hours)
    * long acting β2 agonists (48 hours)
    * ipratropium bromide (12 hours)
    * nasal drops without vasoconstrictors (3 days)
    * DSCG (disodium cromoglycate) (3 days)
    * nedocromil (7 days)
    * nasal drops with vasoconstrictors (7 days)
    * azelastine (14 days)
    * levocabastine (14 days)
    * corticosteroids (30 days)
    * corticosteroids on the site of Prick test (3 months)
    * other investigational drug (3 months)
  * Oral

    * short acting β2 agonists (18 hours)
    * short acting theophylline (24 hours)
    * phenothiazines (48 hours)
    * long acting theophylline (72 hours)
    * anticholinergics (7 days)
    * antihistamines (except astemizole) (7 days)
    * MAO (monoamine oxidase) inhibitors (14 days)
    * corticosteroids (30 days)
    * ketotifen (3 months)
    * imipramine (30 days)
    * astemizole (2 months)
    * other investigational drugs (3 months)
  * Parenteral

    * aminophylline (24 hours)
    * phenothiazines (48 hours)
    * antihistamines (7 days)
    * corticosteroids (30 days)
    * imipramine (30 days)
    * other investigational drugs (3 months)
* Patients under desensitization therapy
* Patients under therapy with antibiotics
* Patients with non compensate endocrine disease
* Patients with atrophic rhinitis
* Patients with rhinitis due to acetylsalicylic acid
* Patients with acute or chronic infectious sinusitis
* Patients with asthma, that need treatment with beta-2 agonists more than twice per week
* Patients with glaucoma
* Patients with history or renal and/or hepatic failure
* Patients with known platelets dysfunction due to any disease or to drugs (purpura thrombocytopenic idiopathic, use of anticoagulants, use of antiplatelets drugs)
* Patients with any oncological disease
* Patients with nasal septal deviation causing alteration of the nasal flux, polyps, anatomic/structural alterations (ex., tumors, leishmaniosis, etc.)
* Patients with any cardiovascular disease
* Patients with arterial hypertension
* Patients requiring halogenates anesthetics
* Patients with diabetes mellitus
* Patients with hyperthyroidism
* Patients with prostatic hypertrophy
* Patients with epilepsy or any other seizure

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2000-05; Primary Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Classification of severity of nasal blockage by Visual Analog Scale (VAS) | at the end of weeks 1, 2, 3, 4
Incidence of laboratory alterations | day 14, 28 and 35
Incidence of premature discontinuations of the study due to adverse events | up to 4 weeks
Incidence and severity of all adverse events | up to 5 weeks

SECONDARY OUTCOMES:
Daily evaluation of the nasal blockage by the patient | daily up to 4 weeks
Classification of the severity of the symptoms by the investigator | at the end of weeks 1, 2, 3, 4
Changes in nasal physical examination | Baseline and at the end of weeks 1, 2, 3, 4
Changes in rhinorrhea symptoms evaluated by investigator | Baseline and at the end of weeks 1, 2, 3, 4
Changes in pruritus symptoms evaluated by investigator | Baseline and at the end of weeks 1, 2, 3, 4
Changes in sneezing symptoms evaluated by investigator | Baseline and at the end of weeks 1, 2, 3, 4
Changes in lacrimation symptoms evaluated by investigator | Baseline and at the end of weeks 1, 2, 3, 4
Changes in rhinorrhea symptoms evaluated by patient using VAS | Baseline and at the end of weeks 1, 2, 3, 4
Changes in pruritus symptoms evaluated by patient using VAS | Baseline and at the end of weeks 1, 2, 3, 4
Changes in sneezing symptoms evaluated by patient using VAS | Baseline and at the end of weeks 1, 2, 3, 4
Changes in lacrimation symptoms evaluated by patient using VAS | Baseline and at the end of weeks 1, 2, 3, 4